CLINICAL TRIAL: NCT03021525
Title: Individualized Perioperative Hemodynamic Goal-directed Therapy in Major Abdominal Surgery (iPEGASUS-trial) - A Multi-center, Prospective, Randomized Trial
Brief Title: Individualized Perioperative Hemodynamic Goal-directed Therapy in Major Abdominal Surgery (iPEGASUS-trial)
Acronym: iPEGASUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University of Giessen (Other); University of Rostock (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 301116
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hemodynamic Instability; Cardiac Output, High; Peroperative Complication
Keywords: Goal-directed therapy; postoperative morbidity; haemodynamic optimisation; individualised medicine; Pulse pressure variation; Cardiac output
MeSH Terms: conditions — Cardiac Output, High; Intraoperative Complications | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Goal Directed Therapy (iGDT) (Experimental): Patients receive fluids and catecholamines following a protocol of individualized parameters achieved by extended hemodynamic monitoring.
  Interventions: Procedure: Individualized Goal Directed Therapy
- Control (Active Comparator): Patients in the control group will be treated according to established basic treatment goals.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Individualized Goal Directed Therapy — The trial intervention period will commence from the induction of anesthesia until 8 hours after surgery, or until discharging from the postoperative intensive or intermediate care unit. All patients in the intervention group receive basic vital sign monitoring. For inotropic support dobutamine, and as vasopressor norepinephrine are drugs of choice. Hemodynamic management is performed according to standard treatment until an arterial line is placed. The signal of the arterial line is then processed either by calibrated or non-calibrated pulse contour analysis for pulse pressure variation (PPV) and cardiac index (CI) measurement. Fluid challenge will be performed by infusion of 500 ml in <15 minute. Choice of fluid in case of indicated fluid loading is determined on basis of the recent guideline for intravasal volume therapy. Patients receive fluids and vasoactive agents following a protocol of individualized parameters regularly achieved by extended hemodynamic monitoring.
  Arms: Individualized Goal Directed Therapy (iGDT)
Procedure: Control Group — Patients in the control group will be treated according to established basic treatment goals (heart rate <100 bpm, mean arterial pressure >65 mmHg, SpO2>94%, and core temperature >36° C). Basic anesthesiological monitoring by five-lead-electrocardiogram, pulse oximetry, non-invasive blood pressure monitoring and capnography is performed in every patient of the control group. Placement of an arterial and central venous line, as well as fluid and catecholamines administration, are at the discretion of the treating clinician.
  Arms: Control

SUMMARY:
To evaluate the impact of perioperative, algorithm driven, hemodynamic therapy based on individualized fluid and cardiac output optimization on postoperative moderate and severe complications in patients undergoing major abdominal surgery including visceral, urological, and gynecological operations.

In the proposed study, hemodynamic therapy is tailored individually to each patient, based on individual preload optimization by the functional parameter "pulse pressure variation (PPV)" and based on an individually titrated goal of cardiac index. The proposed study therefore further develops the concept of hemodynamic goal-directed therapy to individually set goals and is designed to assess its impact on morbidity and mortality.

DETAILED DESCRIPTION:
Postoperative mortality in patients undergoing surgery is on average still 4% in Europe as evaluated recently in a cohort study across 28 European countries and is considered to be even higher in high risk surgery. But besides this significant risk of death, in particular moderate and severe postoperative complications, affecting up to 40% of patients after major surgery, frequently lead to severe reductions of quality of life and cause high healthcare costs in western nations. Perioperative hemodynamic goal-directed optimization is believed to be an integral part to reduce in particular postoperative morbidity significantly and possibly also mortality. Algorithm driven optimization of macrocirculation aiming on best possible oxygen and substrate delivery to end organs and tissues is thought to be the theoretical mechanism of this therapy. A recent large multi-center trial based on such a pragmatic, non-individualized protocol failed to reduce composite morbidity underlining this weak point of this approach. The reason for failing statistically significant improvement of clinical outcome first of all has to be seen in not taking into account individual hemodynamic needs of each single patient. Every patient was hemodynamically treated according to a "one size fits all of maximizing stroke volume" approach. In contrast, a first mono-center trial gave evidence that individualized early goal-directed therapy based on an individually optimized volumetric cardiac preload parameter (global end-diastolic volume) reduces complications and ICU length of stay after cardiac surgery. Further, and even more important, a first multi-center pilot study using a goal-directed algorithm aiming to optimize blood flow oriented on individual cardiac capacities (individualized optimal cardiac index) in major abdominal surgery demonstrated feasibility and a reduction in postoperative complications. This finding needs to be confirmed in a multi-center study that is adequately powered to detect changes in specific complications and in mortality before clinical practice can be changed accordingly. Therefore, the hypothesis of this proposed prospective two arm randomized study is that algorithm driven individualized hemodynamic goal-directed therapy reduces moderate and severe postoperative complications being a massive burden on quality of life and health care costs. The proposed study develops the concept of hemodynamic goal-directed therapy to individually set goals and is designed to assess its impact on morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* To provide high generalizability and representativeness the high number of patients with laparotomy and major surgical trauma is included into this study. - Therefore, open visceral, urological, and gynecological surgery is covered by this study.
* Expected duration of surgery must be ≥ 120 minutes and requirement of volume therapy needs to be expected ≥ 2 liters.
* Risk for any postoperative complications needs to be ≥10% assessed by the ACS (American College of Surgery)- NSQUIP (National Surgical Quality Improvement Program) risk calculator.

Exclusion Criteria:

* Patients <18 years,
* laparoscopic approach,
* patients not having sinus rhythm,
* patients having highly impaired left ventricular function (ejection fraction <30%) or severe aortic valve stenosis (aortic valve area <1 cm2, mean gradient >40 mmHg),
* pregnant women,
* emergency surgeries (surgery required within 24 hours),
* primarily vascular surgery,
* patients suffering from septic shock,
* patients having phaeochromocytoma,
* patients suffering from non-cardiac chest pain,
* refusal of consent,
* patients receiving palliative treatment only (likely to die within 6 months) and patients suffering from acute myocardial ischemia (within 30 days before randomization) are excluded from the study.
* Further, in case that clinicians intended to use cardiac output monitoring for clinical reasons patients should also not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Composite of morbidity and mortality on day 28 | 28 days
  Considering the high relevance for the individual patient and the society, postoperative outcome is most appropriately reflected by a combination of morbidity and mortality. Therefore, the primary endpoint is a composite comprising rate of patients with one or more moderate or severe postoperative complications or death within 28 days post surgery. Moderate and severe postoperative complications are defined on the basis of a consensus statement of an ESA (European Society of Anesthesiology)- ESICM (European Society of Intensive Care Medicine) joint task force on perioperative outcome measures.

SECONDARY OUTCOMES:
Morbidity | Day 1,3,5,7 and 180
  At these days both, number of complications and number of patients having at least one moderate or severe complication, will be assessed in total and for every complication. The additional secondary endpoints including days alive and free of mechanical ventilation at 7 days and 28 days, days alive and free of vasopressor therapy at 7 days and 28 days, days alive and free of renal replacement therapy at 7 days and 28 days, length of ICU and hospital stay further characterize perioperative morbidity and its socioeconomic impacts.
Quality of life after 6 months | Time point of enrolment and on day180
  For assessment of quality of life an interview (personal or by telephone) based on the EQ-5D-5L (EuroQol Research Foundation) questionnaire is performed at the time point of enrolment and 6 months after surgery.
Mortality | Day 180
  Mortality is assessed 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (3):
  - Justus-Liebig-University Giessen, Giessen
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Medicine Rostock, Rostock
- Italy (2):
  - Università degli Studi di Ferrara, Ferrara
  - Università degli Studi di Genova, Genoa
- Spain (2):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari i Politécnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No
To enter a patient into the iPEGASUS trial, research staff at site will log on to a secure web-based randomization system via a link to the respective website and complete the patient's details without individual participant data (name, date of birth etc.) to obtain a unique patient number and allocation to a treatment group. The local main investigator (LMI) will then be informed about patient's enrollment. For correct patient's data follow up only the LMI will set up a list with the possibility to retrace the patient's history. Personalized data will be handled by the LMI according to GCP (good clinical practice) requirements and will be stored separately from the obtained study data. Thereby, data in the eCRF (electronic case report form) itself will not be re-traceable anymore and visible only for the Principal Coordinators (PCs) for data analysis. Data management of the eCRF will be performed by a company specialized in full service study data management.

REFERENCES:
- [Derived] Funcke S, Schmidt G, Bergholz A, Argente Navarro P, Azparren Cabezon G, Barbero-Espinosa S, Diaz-Cambronero O, Edinger F, Garcia-Gregorio N, Habicher M, Klinkmann G, Koch C, Kroker A, Mencke T, Moral Garcia V, Zitzmann A, Lezius S, Pepic A, Sessler DI, Sander M, Haas SA, Reuter DA, Saugel B. Cardiac index-guided therapy to maintain optimised postinduction cardiac index in high-risk patients having major open abdominal surgery: the multicentre randomised iPEGASUS trial. Br J Anaesth. 2024 Aug;133(2):277-287. doi: 10.1016/j.bja.2024.03.040. Epub 2024 May 26. PMID 38797635
- [Derived] Funcke S, Saugel B, Koch C, Schulte D, Zajonz T, Sander M, Gratarola A, Ball L, Pelosi P, Spadaro S, Ragazzi R, Volta CA, Mencke T, Zitzmann A, Neukirch B, Azparren G, Gine M, Moral V, Pinnschmidt HO, Diaz-Cambronero O, Estelles MJA, Velez ME, Montanes MV, Belda J, Soro M, Puig J, Reuter DA, Haas SA. Individualized, perioperative, hemodynamic goal-directed therapy in major abdominal surgery (iPEGASUS trial): study protocol for a randomized controlled trial. Trials. 2018 May 9;19(1):273. doi: 10.1186/s13063-018-2620-9. PMID 29743101